CLINICAL TRIAL: NCT04077125
Title: Minimal Hepatic Encephalopathy is Associated With Increased Cerebral Vascular Resistance. a Transcranial Doppler Ultrasound Study
Brief Title: Transcranial Doppler Ultrasound and Minimal Hepatic Encephalopathy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Francesca Ponziani, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1712
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Minimal Hepatic Encephalopathy
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cirrhosis no MHE: Patients with liver cirrhosis without signs of minimal hepatic encephalopathy
- Cirrhosis MHE: Patients with liver cirrhosis with minimal hepatic encephalopathy
  Interventions: Drug: Rifaximin
- Controls: Healhty subjects

INTERVENTIONS:
Drug: Rifaximin — to investigate changes in cerebral, splanchnic hemodynamics and endothelial function in cirrhotic patients with MHE after 15 days of rifaximin therapy (1200 mg/d)
  Groups: Cirrhosis MHE

SUMMARY:
Minimal hepatic encephalopathy (MHE) is a subclinical complication of liver cirrhosis with a relevant social impact. Thus, there is urgent need to implement easy to use diagnostic tools for the early identification of affected patients.

This study was aimed to investigate cerebral blood flow, systemic hemodynamics as well as endothelial function of cirrhotic patients with MHE, and to verify their change after treatment with rifaximin.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of liver cirrhosis on the basis of clinical, laboratory and ultrasound findings

Exclusion Criteria:

* active alcohol abuse (excessive alcohol intake stopped more than 6 months before the enrollment);
* chronic pulmonary diseases; ongoing infections; cerebrovascular diseases; primary or secondary cerebral neoplasm; primary liver neoplasm; heart function failure; chronic kidney disease; peripheral vascular disease; treatment with rifaximin or systemic antibiotics in the previous 15 days;
* smoking habit;
* grade 1 or overt hepatic encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All cirrhotic patients evaluated at the Department of Internal Medicine, Gastroenterology and Hepatology of the Fondazione Policlinico A. Gemelli in Rome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Quantification of middle cerebral artery resistive index | baseline
  Quantification of middle cerebral artery resistive index by Doppler ultrasound in patients with liver cirrhosis with or without MHE
Quantification of middle cerebral artery pulsatility index | baseline
  Quantification of middle cerebral artery pulsatility index by Doppler ultrasound in patients with liver cirrhosis with or without MHE
Quantification of posterior cerebral artery resistive index | baseline
  Quantification of posterior cerebral artery resistive index by Doppler ultrasound in patients with liver cirrhosis with or without MHE
Quantification of posterior cerebral artery pulsatility index | baseline
  Quantification of posterior cerebral artery pulsatility index by Doppler ultrasound in patients with liver cirrhosis with or without MHE
Change in middle cerebral artery resistive index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Variation of middle cerebral artery resistive index measured by Doppler ultrasound after treatment with rifaximin 1200 mg/d for 15 days in patients with liver cirrhosis and MHE
Change in middle cerebral artery pulsatility index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Variation of middle cerebral artery pulsatility index measured by Doppler ultrasound after treatment with rifaximin 1200 mg/d for 15 days in patients with liver cirrhosis and MHE
Change in posterior cerebral artery resistive index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Variation of posterior cerebral artery resistive index measured by Doppler ultrasound after treatment with rifaximin 1200 mg/d for 15 days in patients with liver cirrhosis and MHE
Change in posterior cerebral artery pulsatility index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Variation of posterior cerebral artery pulsatility index measured by Doppler ultrasound after treatment with rifaximin 1200 mg/d for 15 days in patients with liver cirrhosis and MHE

SECONDARY OUTCOMES:
Comparison of renal artery resistive index of cirrhotic patients with MHE compared to those without | baseline
  Comparison of renal artery resistive index measured by Doppler ultrasound of cirrhotic patients with MHE and those without
Comparison of splenic artery resistive index of cirrhotic patients with MHE compared to those without | baseline
  Comparison of splenic artery resistive index measured by Doppler ultrasound of cirrhotic patients with MHE and those without
Comparison of flow mediated dilation of cirrhotic patients with MHE compared to those without | baseline
  Comparison of endothelial function (flow mediated dilation measured by Doppler ultrasound) of cirrhotic patients with MHE and those without
Change in renal artery resistive index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Change in renal artery resistive index measured by Doppler ultrasound in patients with liver cirrhosis and MHE after treatment with rifaximin 1200 mg/d for 15 days
Change in splenic artery resistive index after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Change in splenic artery resistive index measured by Doppler ultrasound in patients with liver cirrhosis and MHE after treatment with rifaximin 1200 mg/d for 15 days
Change in flow mediated dilation after treatment with rifaximin | at the end of rifaximin treatment (15 days)
  Change in endothelial function (flow mediated dilation measured by Doppler ultrasound) in patients with liver cirrhosis and MHE after treatment with rifaximin 1200 mg/d for 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No